CLINICAL TRIAL: NCT04232540
Title: Establishing Novel Antiretroviral Imaging for Hair to Elucidate Non-Adherence (ENLIGHTEN)
Acronym: ENLIGHTEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-3360; R01AI122319 (NIH); 122319 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Medication Adherence
Keywords: HIV infection; Medication Adherence; Hair; Dolutegravir; Emtricitabine; Antiretrovirals
MeSH Terms: conditions — Medication Adherence; HIV Infections

STUDY DESIGN:
Intervention Model Description: Dual Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Patient participants (Experimental): Patient and provider will view and discuss results of the MedViewer test.
  Interventions: Device: MedViewer report
- Provider participants (Experimental): Patient and provider will view and discuss results of the MedViewer test.
  Interventions: Device: MedViewer report

INTERVENTIONS:
Device: MedViewer report — Results from the analysis of hair samples performed using the MedViewer

SUMMARY:
This is a pilot study to assess the feasibility, acceptability and appropriateness of delivery of the investigational "MedViewer" intervention in adult patients living with HIV who have been prescribed antiretroviral (ARV) medications. The Medviewer uses Infra-red (IR) matrix-assisted laser desorption electrospray ionization (MALDESI) technology for mass spectrometry imaging (MSI) to analyze patient hair samples to provide information on ARV adherence in real-time.

The study has two different groups of participants: the patients, and their clinician providers.

DETAILED DESCRIPTION:
This study is part of a larger research program that is investigating a novel non-invasive approach to rapidly quantify ARV concentrations and provide evidence of drug ingestion. The ultimate goal is to provide clinicians and patients feedback on ARV adherence. Infra-red (IR) matrix-assisted laser desorption electrospray ionization (MALDESI) technology for mass spectrometry imaging (MSI) is used to visualize and quantify ARV concentrations in hair. The IR-MALDESI MSI has been labeled the "MedViewer".

Patient participants will be scheduled for the sampling visit to correspond with their next appointment at the University of North Carolina (UNC) Infectious Disease (ID) clinic. Patient participants will be asked to arrive to their clinic appointment at least two hours prior to the scheduled time to be consented and enrolled. If eligible and enrolled in the study, patient participants will have a small hair sample (5 strands) plucked from a discrete location on the back of their head. Patient participants will also have a small blood sample collected. The results from the MedViewer test will be provided to both the patient and their provider, in order to facilitate a discussion around medication adherence. After receiving the results, all participants will complete a brief questionnaire about their experience with the MedViewer.

As this is a feasibility study, results from the Medviewer test will not be used to make clinical decisions related to care.

Major changes after the start of enrollment:

1. Removed the term "real-time" throughout the document-Pertinent feasibility endpoints now use "delivery of the report to the designated research staff member within 2 hours of initiation of hair processing" rather than "…within 2 hours of hair sample collection"
2. Removed mitra sampling for the remaining 15 participants in cohort A. Now stated as "blood sample will be collected for 10 participants in Group A and a subset of participants in Group B." After Mitra is analyzed for the first 10 participants in Group B, we will reevaluate to determine if additional samples are needed to validate hair samples.
3. V1 and V2 study activities will be conducted virtually (except hair collection and in-person patient provider clinic visits) to minimize in-person contact. Consent and screening will be conducted virtually using videoconferencing via zoom on computer, tablet or phone. All questionnaires (patient baseline, patient post-visit, patient endline, provider baseline, provider post-visit, and provider endline) will be conducted virtually through REDCap (emailed to participant or verbally administered via phone or videoconferencing). Hair collection will be conducted by research staff at remote locations to limit time in clinic. Implementation of the intervention will now be allowed in the setting of telehealth clinical visits between patient and provider in addition to in-person clinical visits. MedViewer reports will be sent to providers via secure email. All remaining V2s will be conducted virtually. Hair and blood samples will not be collected.
4. Consenting will take place up to 3 days before scheduled clinic appointment with provider. Hair sample will be collected by research staff at a remote location in the 3 days between consent and the scheduled provider visit. MedViewer report will be discussed between patient and provider (or patient and pharmacist, if needed) within 4 weeks of hair sample collection.
5. Interviewer-administered portions of the baseline questionnaire have been modified. Health Literacy measure (Newest Vital Sign) removed. ART adherence Visual Analog Scale modified to allow for remote self-administration.
6. Maximum duration on study extended by 6 months for providers (increased from 10 to 16 months). Provider sample size range reduced (from 20-30 to 16-30)

These changes were implemented on November 5, 2020 in a Letter of Amendment (LOA) to ENLIGHTEN Protocol Version 2. The LOA detailed changes made to the protocol due to the COVID-19 Pandemic.

ELIGIBILITY:
Inclusion Criteria:

Patient participants:

* Documentation of HIV-1 infection by means of any one of the following:

  1. Documentation of HIV diagnosis in the medical record by a licensed health care provider;
  2. OR HIV-1 RNA detection by a licensed HIV-1 RNA test demonstrating >1000 RNA copies/mL;
  3. OR any licensed HIV screening antibody and/or HIV antibody/antigen combination test confirmed by a second licensed HIV test such as a HIV-1 Western blot confirmation or HIV rapid Multispot antibody differentiation test.
* At least 18 years of age on the day of consent.
* Documentation of HIV viral loads over 2-year period prior to screening.
* Has been a patient at the UNC ID clinic for at least 90 consecutive days prior to the date of enrollment in the study (i.e. attended first appointment at the UNC ID Clinic at least 90 days prior to the date of enrollment in the study).
* Has attended at least one HIV appointment at the UNC ID clinic within the 365 days prior to the date of enrollment in the study.
* Has been prescribed one of the ARV medications eligible in this study (Dolutegravir, Emtricitabine) by a UNC provider for at least 90 days prior to the date of enrollment in the study.
* Has an HIV appointment scheduled at the UNC ID clinic during the enrollment period of the study with a medical provider enrolled in the study.
* Evidence of a personally signed and dated informed consent form indicating that the participant has been informed of all pertinent aspects of the study.
* Has stated willingness and availability to comply with all study procedures for the duration of the study.
* Literate in English.
* Has at least 1.0 cm of natural caput hair.
* As enrollment will occur in a stratified manner based on 2 viral load strata, (n = 25 for patients with undetectable viral loads, n = 25 for those with detectable viral loads), once a stratum quota is reached, patients whose viral loads fall within that stratum will not be eligible to participate in the study.

Provider participants:

* Medical provider (including, but not limited to: attending physician, ID fellow, nurse practitioner, physician assistant, or a designated HIV Care pharmacist) for UNC ID clinic patients living with HIV.
* Provides medical care for patients at the UNC ID clinic at least one half-day per week (i.e. 4 hours per week).
* Evidence of a personally signed and dated informed consent form indicating that the participant has been informed of all pertinent aspects of the study.
* Has stated willingness and availability to comply with all study procedures for the duration of the study.

Exclusion Criteria:

Patient participants:

* Previous participation in the study UNC 11530- Formative Sub-Study for Novel Mass Spectrometry Imaging Methods to Quantify Antiretroviral Adherence.
* Deemed, by medical provider in UNC ID clinic, too ill, or other relevant reason, to participate in the study.
* Prior history of clinically significant alteration of the gastrointestinal system or drug absorption capability, including but not limited to: gastrectomy, total colectomy
* Any chemical hair treatment with dye, bleach, or relaxers within the past 4 weeks prior to sampling

Provider participants:

* Not willing or able to participate in any of the provider training sessions for this study or any form of make-up training session with research team.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Kashuba, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Response to individual request for raw data. Any resulting publication from this proposal will include the principle investigator or a co-investigator listed on the application as corresponding author. Raw de-identified datasets will be shared with requesting scientists at the discretion of principle investigator to foster scientific openness in an ethical and responsible manner.
Supporting Information: CSR
Time Frame: Upon acceptance of final manuscript for publication for an indefinite time period
Access Criteria: Before data will be shared, a data use agreement will be put in place in accordance with local regulations. The requestor will need to obtain appropriate ethics approval.
URL: http://unc.edu

REFERENCES:
- [Derived] Golin CE, Rosen EP, Ferguson EG, Perry NR, Poliseno AJ, Munson AJ, Davis A, Hill LM, Keys J, White NR, Farel CE, Kashuba A. Feasibility, Acceptability and Appropriateness of MedViewer: A Novel Hair-Based Antiretroviral Real-Time Clinical Monitoring Tool Providing Adherence Feedback to Patients and Their Providers. AIDS Behav. 2023 Dec;27(12):3886-3904. doi: 10.1007/s10461-023-04104-1. Epub 2023 Jul 26. PMID 37493932
- [Derived] Poliseno A, Ferguson E, Perry R, Munson A, Davis A, Hill L, Keys J, White N, Farel C, Gay C, Golin C, Rosen E, Kashuba A. Establishing Novel Antiretroviral Imaging for Hair to Elucidate Nonadherence: Protocol for a Single-Arm Cross-sectional Study. JMIR Res Protoc. 2023 Apr 21;12:e41188. doi: 10.2196/41188. PMID 37083754

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Participants | Provider Participants
Started | 37 | 20
Received MedViewer (The MedViewer report was received as planned if results were: (1) delivered to the research team member within 2 hours of initiation of hair sample processing; and (2) discussed between the patient and provider/pharmacist during their clinic visit.) | 34 | 16
Completed In-Depth Interview | 24 | 14
Completed | 36 | 20
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Participants | Provider Participants | Total
Number analyzed (Participants) | 37 | 20 | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [37 to 57] | 44.5 [37 to 53] | 49 [37 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 23 | 7 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 35 | 20 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 1 | 22
  White | 13 | 17 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patient Participants That Received a MedViewer Report as Planned
Description: Patient participants received their MedViewer report as planned if: (1) they had results delivered to the research team member within 2 hours of initiation of hair sample processing; and (2) discussed results with a provider participant during their clinic visit. The percent of patient participants that received the MedViewer report as planned is reported.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit
Population: All patient participants were included in the analysis.
Measure: Number; unit: percentage of patient participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 37
percentage of patient participants | 91.9

2. Primary Outcome: Percent of Contacted Patients That Were Eligible for a Screening Visit and Agreed to Participate in the Study
Description: Contacted patients were deemed eligible for a screening visit using a pre-screening questionnaire and provided documented informed consent to participate in the study. The percent of all contacted eligible patients that agreed to participate in study is reported. Per study protocol, this outcome is not measured in providers.
Time Frame: Visit 1 (Day 1) before patient participant clinic visit
Population: All patients that were contacted and deemed eligible for study were included in the analysis.
Measure: Number; unit: percentage of contacted patients
Arm/Group | Patient Participants
Number analyzed (Participants) | 75
percentage of contacted patients | 49.3

3. Primary Outcome: Percent of Patient Participants That Were Satisfied With Their Discussion With a Provider Participant About Antiretroviral (ART) Adherence Using the MedViewer Report
Description: Patient participants were asked to rate their satisfaction with the MedViewer report for promoting a productive discussion of ART adherence with a provider participant. Satisfaction was rated on a rated on a 5-point scale (1="very unsatisfied" to 5="very satisfied"), with higher scores being more favorable. The percent of patient participants reporting 4 or greater (4="somewhat satisfied" or 5="very satisfied") on this scale as was calculated.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit
Population: Patient participants that received a MedViewer report and discussed the report with a provider participant as planned were included in the analysis.
Measure: Number; unit: percentage of patient participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 34
percentage of patient participants | 100

4. Primary Outcome: Percent of Patient Participants for Whom Provider Participants Reported the MedViewer Report as Being Useful for Promoting a Productive Antiretroviral (ART) Adherence Discussion
Description: For each of patient participant, provider participants were asked to rate the usefulness of the MedViewer report in promoting a productive discussion with the patient participant about ART adherence using a 5-point scale (1="not at all useful" to 5="extremely useful"), with a higher score being more favorable. The percent of patient participants with provider participants reporting 4 or greater (4="very useful" or 5="extremely useful") on this scale as was calculated.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit
Population: as for outcome 3
Measure: Number; unit: percentage of patient participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 34
percentage of patient participants | 58.8

5. Secondary Outcome: Among Patient Participants That Did Dot Receive a MedViewer Report, Percent of Patient Participants That Did Not Receive the MedViewer for a Given Reason or Reasons
Description: Reasons for patient participants' non-receipt of MedViewer report were only assessed for the subset of patient participants for whom non-receipt was reported. Reasons for non-receipt were assessed by provider participants for each patient participant after their scheduled visit using a single multiple-choice, multiple-answer question. The percent of patient participants for whom a reason or combination of reasons for non-receipt is reported.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit
Population: Patient participants that did not receive and/or discuss a MedViewer report with a provider participant as planned were included in the analysis.
Measure: Number; unit: percentage of patient participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 3
percentage of patient participants
  Technical Difficulties, Provider Did Not Think It Was Beneficial to Show Report to Patient | 33.3
  No Time to Show Report, Did Not Receive Report Before Visit | 33.3
  Patient Had More Pressing Medical Issues | 0
  Other | 33.3

6. Secondary Outcome: Mean Hours From Patient Participant Hair Sample Processing Initiation to MedViewer Report Delivery to Designated Research Staff Member
Description: For each patient participant, the number of hours elapsed from the time of initiation of hair processing in the lab (Time 1) to the time of results delivery to designated research staff member (Time 2) was calculated, and a population mean was determined.
Time Frame: Time 1 to Time 2 prior to or on Visit 1 (Day 1)
Population: All patient participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Patient Participants
Number analyzed (Participants) | 37
hours | 1.80 (0.414)

7. Secondary Outcome: Percent of Participants Reporting a High Likelihood of Future MedViewer Report Use
Description: The 4-point scale measuring the likelihood of future MedViewer report use ranged from 1="definitely would not" to 4="definitely would", with a higher score being more favorable. The percent of participants that scored 3 or greater on the likelihood of future MedViewer use scale (3="probably would" or "4="definitely would") was calculated.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit for patient participants, end line visit for provider participants
Population: All patient participants were included in the analysis. Only provider participants that saw patient participants were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Patient Participants | Provider Participants
Number analyzed (Participants) | 37 | 16
percentage of participants | 97.2 | 100

8. Secondary Outcome: Percent of Patient Participants Reporting High Comprehension of the MedViewer Report
Description: Patient participants were asked to rate their comprehension of the information presented in the MedViewer report using a 4-point scale (1="very difficult to understand" to 4="very easy to understand"), with a higher score being more favorable. The percent of patient participants reporting 3 or greater on this scale (3="somewhat easy to understand" or 4="very easy to understand") was calculated.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit
Population: as for outcome 3
Measure: Number; unit: percentage of patient participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 34
percentage of patient participants | 97.1

9. Secondary Outcome: Percent of Patient Participants Reported by Provider Participants as Having High Comprehension of the MedViewer Report
Description: Provider participants were asked to rate each of patient participant's comprehension of the information presented in the MedViewer report using a 5-point scale (1="understood not at all well" to 5="understood excellently"), with a higher score being more favorable. The percent of patient participants with provider participants reporting 4 or greater (4="understood very well" or 5="understood excellently") on this scale as was calculated.
Time Frame: Visit 1 (Day 1) after patient participant clinic visit
Population: as for outcome 3
Measure: Number; unit: percentage of patient participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 34
percentage of patient participants | 73.5

10. Secondary Outcome: Mean Usefulness Score for the MedViewer Report to Promote ART (Antiretroviral) Adherence
Description: Participants were asked to rate their perceived usefulness of the MedViewer report for promoting ART adherence. Usefulness was rated on a rated on a 5-point scale (1="not at all useful" to 5="extremely useful"), with higher scores being more favorable. A mean usefulness score was calculated for each participant.
Time Frame: as for outcome 7
Population: Patient participants that discussed the MedViewer as planned were included in the analysis. Provider participants that saw patient participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Participants | Provider Participants
Number analyzed (Participants) | 34 | 16
score on a scale | 4.2 (0.999) | 4.00 (1.033)

11. Secondary Outcome: Percent of Participants That Reported a Positive Change in the Patient-provider Relationship After Using the MedViewer Report
Description: Participants were asked to rate the comparative satisfaction with patient participant-provider participant discussions during the MedViewer visits as compared to typical visits. Patient participants were asked this question after Visit 1, while provider participants were asked this question at their end line visit. Change in relationship was rated on 5-point scale (1="much less satisfied than usual" to 5="much more satisfied than usual"), with a higher score being more favorable. The percent of participants reporting 4 or greater on this scale (4="somewhat more satisfied than usual" or 5="much more satisfied than usual") was calculated.
Time Frame: as for outcome 7
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Patient Participants | Provider Participants
Number analyzed (Participants) | 34 | 16
percentage of participants | 88.2 | 50.0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the interval from hair sample collection to end line visit, up to a total of 28 days.
Arm/Group | Patient Participants | Provider Participants
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/20
Other Adverse Events (participants affected / at risk) | 0/37 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04232540/Prot_SAP_ICF_000.pdf